CLINICAL TRIAL: NCT05092529
Title: The Psychological Impact of Surviving an Intensive Care Admission Due to Coronavirus Disease 2019 (COVID-19) on Patients in the United Kingdom
Brief Title: Psychological Impact of COVID-19 on Intensive Care Survivors
Acronym: PIM-COVID
Status: Completed | Type: Observational
Sponsor: Royal Liverpool University Hospital (Other Government)
Responsible Party: Principal Investigator, Alicia Waite, Postdoctoral Clinical Research Fellow, Royal Liverpool University Hospital
Other Study IDs: SP0316; IRAS 282400 (Registry Identifier: IRAS); NIHR CPMS 47545 (Registry Identifier: NIHR CPMS)
Record Dates: First submitted 2021-10-18; First posted 2021-10-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Psychological Distress; Depression; Anxiety; Post-traumatic Stress Disorder; Post Intensive Care Syndrome
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychological distress is commonly experienced by survivors of an intensive care admission, including patients treated during previous pandemics. Whilst data emerges about the short-term impact of COVID-19 on patients and healthcare systems, the long term impact remains unclear.

The purpose of this trainee-led, multi-centre longitudinal study is to assess the short- and long-term psychological impact on patients who have survived an admission to intensive care due to COVID-19, and identify possible predictors of anxiety, depression and trauma symptoms in this patient group.

DETAILED DESCRIPTION:
The primary objective is to identify the proportion of patients surviving an admission to intensive care due to COVID-19 who experience anxiety, depression and/or trauma symptoms in the 6 months post discharge.

Whilst the secondary objectives are to identify demographic, clinical, physical and/or psychosocial predictors of depression, anxiety and/or trauma symptoms at 3-, 6- and 12-months post discharge from ICU. And to assess the feasibility of using a self-reported online questionnaire to assess anxiety, depression and/or trauma symptoms in patients following ICU admission.

An amendment was approved by the East Midlands - Derby Research Ethics Committee on 17 March 2022, to conduct three sub-studies:

1. Semi-structured interviews - to explore the experiences of critical care survivors following COVID-19 infection during their recovery phase, including perceptions about the care received and support available to them.
2. Survey of follow-up services offered to ICU survivors - to assess geographical differences in the availability and structure of follow-up services offered to patients with critical COVID-19 after hospital discharge.
3. Survey of study team members - to gain feedback from the study team members on their involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Survival to intensive care / high dependency unit discharge following an admission of ≥24 hours
* Treated for COVID-19

Exclusion Criteria:

* Unable to complete questionnaires
* Unable or unwilling to consent
* Unable to speak, understand or communicate in English
* Patients with diagnosed, pre-existing cognitive impairment (at the time of ICU admission)
* Patients without a fixed abode, at which postal questionnaires might be received, and who have no access to a personal email address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care survivors
Sampling Method: Non-Probability Sample
Enrollment: 1620 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Anxiety | 6 months post intensive care unit (ICU) discharge
  Hospital Anxiety and Depression Scale (HADS) where a score of 0-7= normal, 8-10= borderline abnormal (borderline case), 11-21= abnormal (case).
Depression | 6 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS) where a score of 0-7= normal, 8-10= borderline abnormal (borderline case), 11-21= abnormal (case).
Symptoms of trauma | 6 months post ICU discharge
  Impact of Event Scale-6 (IES-6) where the mean score ranges between 0 and 4 and the cut off score is 1.75.

SECONDARY OUTCOMES:
Anxiety | 3 and/or 12 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS) where a score of 0-7= normal, 8-10= borderline abnormal (borderline case), 11-21= abnormal (case).
Depression | 3 and/or 12 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS) where a score of 0-7= normal, 8-10= borderline abnormal (borderline case), 11-21= abnormal (case).
Symptoms of trauma | 3 and/or 12 months post ICU discharge
  Impact of Event Scale-6 (IES-6) where the mean score ranges between 0 and 4 and the cut off score is 1.75.
Metacognitive beliefs and processes | 3, 6 and/or 12 months post ICU discharge
  Cognitive Attentional Syndrome Scale-1 (Revised; CAS-1R), which is a 10-item measure with responses scaled from 0%-100%, which are summed to produce a total score. Higher scores indicate greater conviction in metacognitive beliefs and greater use of maladaptive coping strategies to manage distress.
Health-related quality of life | 3, 6 and/or 12 months post ICU discharge
  EuroQol 5-dimension, 5-level questionnaire (EQ-5D-5L) comprises health status measures (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) divided into five levels of perceived problems and a visual analogue scale of health status ranging from 0-100.
Feasibility of using self-reported questionnaire to assess psychological outcomes in ICU survivors with COVID-19 | Study duration, up to 1 year
  Response rate to invitations to participate/questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia AC Waite, Principal Investigator — Royal Liverpool University Hospital; Ingeborg D Welters, Principal Investigator — University of Liverpool
Locations (50):
- United Kingdom (50):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Barnsley Hospital, Barnsley, England
  - Basildon Hospital, Basildon, England
  - Bedford Hospital, Bedford, England
  - Royal Blackburn Hospital, Blackburn, England
  - Pilgrim Hospital, Boston, England
  - Royal Papworth Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Countess of Chester Hospital, Chester, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Colchester Hospital, Colchester, England
  - Leighton Hospital, Crewe, England
  - Wonford Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Ipswich Hospital, Ipswich, England
  - Kingston Hospital, Kingston upon Thames, England
  - Lincoln County Hospital, Lincoln, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Lewisham and Greenwich Hospitals, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Maidstone Hospital, Maidstone, England
  - James Cook University Hospital, Middlesbrough, England
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, England
  - Newcastle upon Tyne Hospitals Foundation Trust, Newcastle upon Tyne, England
  - Northampton General Hospital, Northampton, England
  - Nottingham University Hospitals, Nottingham, England
  - Royal Oldham Hospital, Oldham, England
  - Derriford Hospital, Plymouth, England
  - Whiston Hospital, Prescot, England
  - Rotherham General Hospital, Rotherham, England
  - Tunbridge Wells Hospital, Royal Tunbridge Wells, England
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, England
  - Lister Hospital, Stevenage, England
  - King's Mill Hospital, Sutton in Ashfield, England
  - Musgrove Park Hospital, Taunton, England
  - Pinderfields General Hospital, Wakefield, England
  - Watford General Hospital, Watford, England
  - Royal Albert Edward Infirmary, Wigan, England
  - Ulster Hospital, Belfast, Northern Ireland
  - Forth Valley Royal Hospital, Larbert, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Royal Glamorgan Hospital, Pont-y-clun, Wales
  - Morriston Hospital, Swansea, Wales
  - North Middlesex University Hospital, London
  - Southend University Hospital, London
  - Manchester Royal Infirmary, Manchester
  - North Manchester General Hospital, Manchester
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford

IPD SHARING:
Plan to Share IPD: Undecided
Upon the conclusion of the study, the dataset may be made available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Waite AAC, Johnston BW, Boyle AJ, Cherry MG, Fisher P, Brown SL, Jones C, Williams K, Welters ID. PIM-COVID study: protocol for a multicentre, longitudinal study measuring the psychological impact of surviving an intensive care admission due to COVID-19 on patients in the UK. BMJ Open. 2023 Sep 27;13(9):e071730. doi: 10.1136/bmjopen-2023-071730. PMID 37758678
- See also: Trainee Research in Intensive Care Network website — http://tricnetwork.co.uk

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT05092529/Prot_SAP_ICF_002.pdf